CLINICAL TRIAL: NCT02422979
Title: A Phase 1/2a Multicenter, Open-Label, Dose-Escalation, Combination Study of RM-1929 and Photoimmunotherapy in Patients With Recurrent Head and Neck Cancer, Who in the Opinion of Their Physician, Cannot Be Satisfactorily Treated With Surgery, Radiation or Platinum Chemotherapy
Brief Title: Study of RM-1929 and Photoimmunotherapy in Patients With Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rakuten Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RM-1929/101
Record Dates: First submitted 2015-04-03; First posted 2015-04-22 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Recurrent Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- PART 1 - Cohort 1 (Experimental): 3-6 patients
  Interventions: Combination Product: PIT: 50 J/cm^2 for superficial lesions or 100 J/cm for interstitial lesions and Drug RM-1929: 160 mg/m^2
- PART 1 - Cohort 2 (Experimental): 3-6 patients
  Interventions: Combination Product: PIT: 50 J/cm^2 for superficial lesions or 100 J/cm for interstitial lesions and Drug RM-1929: 320 mg/m^2
- PART 1 - Cohort 3 (Experimental): 3-6 patients
  Interventions: Combination Product: PIT: 50 J/cm^2 for superficial lesions or 100 J/cm for interstitial lesions and Drug RM-1929: 640 mg/m^2
- PART 2 - Cohort 1 (Experimental): Number of patients depend on Part 1
  Interventions: Combination Product: PIT: 75 J/cm^2 for superficial lesions or 150 J/cm for interstitial lesions and Drug RM-1929: 640mg/m^2
- PART 2 - Cohort 2 (Experimental): Number of patients depend on Part 1
  Interventions: Combination Product: PIT: 100 J/cm^2 for superficial lesions or 200 J/cm for interstitial lesions and Drug RM-1929: 640mg/m^2
- PART 3 (Experimental): Up to 30 patients
  Interventions: Combination Product: PIT: 50 J/cm^2 for superficial lesions or 100 J/cm for interstitial lesions and Drug RM-1929: 640mg/m^2

INTERVENTIONS:
Combination Product: PIT: 50 J/cm^2 for superficial lesions or 100 J/cm for interstitial lesions and Drug RM-1929: 160 mg/m^2
  Arms: PART 1 - Cohort 1
Combination Product: PIT: 50 J/cm^2 for superficial lesions or 100 J/cm for interstitial lesions and Drug RM-1929: 320 mg/m^2
  Arms: PART 1 - Cohort 2
Combination Product: PIT: 50 J/cm^2 for superficial lesions or 100 J/cm for interstitial lesions and Drug RM-1929: 640 mg/m^2
  Arms: PART 1 - Cohort 3
Combination Product: PIT: 75 J/cm^2 for superficial lesions or 150 J/cm for interstitial lesions and Drug RM-1929: 640mg/m^2
  Arms: PART 2 - Cohort 1
Combination Product: PIT: 100 J/cm^2 for superficial lesions or 200 J/cm for interstitial lesions and Drug RM-1929: 640mg/m^2
  Arms: PART 2 - Cohort 2
Combination Product: PIT: 50 J/cm^2 for superficial lesions or 100 J/cm for interstitial lesions and Drug RM-1929: 640mg/m^2
  Arms: PART 3

SUMMARY:
This is a two-part clinical study of patients with recurrent Head and Neck Cancer (HNC), who in the opinion of their physician, cannot be satisfactorily treated with surgery, radiation or platinum chemotherapy. The purpose of the study is to determine the safety and anti-cancer activity of various doses and repeated cycles of the experimental treatment using the study drug RM-1929 and fixed amounts of red light applied at the tumor site to activate the pharmacodynamics of the drug.

The part 1 of the study has been completed and consisted in a single cycle, 3+3 dose escalation safety study of the experimental drug RM-1929 using a fixed amount of 690 nm red light. The part 1 was designed to determine the safety of the treatment as set by the maximal feasible dose or the maximal tolerable dose of RM-1929. From the part 1 results, the maximal feasible dose of RM-1929 was determined.

The part 2 of the study is currently ongoing and it is evaluating the safety and anticancer efficacy of up to four repeated treatments of Photoimmunotherapy with RM-1929 at the maximal feasible dose of RM-1929 activated with a fixed amount of red light.

DETAILED DESCRIPTION:
Photoimmunotherapy (PIT) is a new cancer targeted technology invented at the National Cancer Institute, USA. This clinical study evaluates the treatment of the experimental drug RM-1929 with Photoimmunotherapy (PIT).

The experimental drug, RM-1929, is a parental formulation consisting of a chemical conjugate of the dye IR700 with the FDA approved antibody, Erbitux® (Cetuximab), that targets EGFR receptors (EGFR is a cancer expressed protein, a cancer antigen). EGFR is highly expressed in squamous cell carcinomas of the head and neck (HNSCC). It is expected that systemic administration of RM-1929 will lead to tumor accumulation and binding to EGFR expressed at cancer cells. It is expected that treatment with RM-1929 and Photoimmunotherapy can lead to the selective destruction of the HNSCC cancer cells and provide an effective therapy to manage the disease.

The treatment using RM-1929 with Photoimmunotherapy requires two steps:

(i) the administration by infusion of the drug RM-1929 targeting the cancer protein EGFR

AND

(ii) the illumination of the tumor with red light (690 nm) using sufficient energy to activate the drug and induce cancer cell killing.

Light illumination is applied at 24 h post drug infusion to enable sufficient time for the drug to distribute in the tumor after administration. Cell killing occurs only at cancer cells expressing the protein EGFR that is bound to the drug RM-1929. The requirement of binding of the drug to EGFR of cancer cells enables the selective destruction of cancer cells with minimum damage of healthy tissue surrounding the tumor cells. Preclinical pharmacology demonstrated that light-induced activation of RM-1929 elicits rapid tumor destruction of human cancer xenografts implanted in mice and that the treatment is cancer specific.

The Part 1 study has been completed and consisted of a single cycle 3+3 dose escalation study of RM-1929 to determine the safety of the treatment and the maximal feasible dose of RM-1929. From the part 1 of this study, the maximal feasible dose for treatment with RM-1929 was selected. The currently ongoing Part 2 of the clinical study is evaluating the safety and anti-cancer activity of up to 4 repeat treatment cycles of Photoimmunotherapy with RM-1929.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria to be eligible for study participation:

1. Patients with recurrent squamous carcinoma of the Head and Neck, who in the opinion of their treating physician, cannot be satisfactorily treated with surgery, radiation, or platinum chemotherapy. Diagnosis must be confirmed by biopsy and histopathology.
2. Patient must have received prior systemic platinum-based chemotherapy for treatment of their head and neck cancer, unless in the opinion of the medical oncologist, the use of platinum-based chemotherapy is contraindicated or not recommended, e.g., renal impairment, allergy to platinum compounds, age, liver disease, myelosuppression, neuropathy, hearing loss, etc.
3. Patients must have life expectancy > 6 months based on investigator judgment.
4. Male or female patients at least 18 years old. Female patients must not be pregnant or breast feeding and must be practicing a medically acceptable form of birth control, be sterile, or post-menopausal. Females of childbearing potential (FCBP) is defined as premenopausal women capable of becoming pregnant. This includes women who are post-menopausal for at least 12 months after the last menses. FCBP must agree to use a medically acceptable form of birth control during the study and for at least 6 months after discontinuation of Erbitux® or study medication. Females must agree not to breast feed during the study and for at least two months after discontinuation of Erbitux® or study medication. Male patients should be using a double barrier protection method that is a medically acceptable form of birth control during the study or be sterile.
5. Patients must have an ECOG score of 0 - 2.
6. Patient must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

Patients with any of the following will be excluded from participation in the study:

1. Patients with a history of significant Erbitux infusion reactions (≥ Grade 3).
2. Patients on chemotherapy or Erbitux® therapy or radiation therapy within 4 weeks of enrollment.
3. Tumor invading a major blood vessel (such as the carotid artery) unless the vessel has been embolized, stented or surgically ligated to prevent hemorrhage.
4. Tumor is not clearly shown on a CT scan or clinically measurable.
5. Location and extension of the tumor precludes an effective PIT.
6. Patients with impaired hepatic function (ALP (hepatic), AST and/or ALT >3 times the upper normal limits, or total serum bilirubin > 2 mg/dL.
7. Patients with impairment of renal function (serum creatinine >2 mg/dL).
8. Unwilling or unable to follow protocol requirements.
9. Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive study drug.
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
11. Patient requires examinations or treatments within 4 weeks after study drug administration where they would be exposed to significant light, e.g., eye examinations, surgical procedures, endoscopy, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Part I: Maximum Tolerated Dose (MTD) or Maximum Feasible Dose (MFD) of RM-1929, whichever is lowest | 1 month
  Determine the MTD or MFD of RM-1929
Part I: Adverse Event profile for each drug dose of RM-1929 | 1 month
  Assessment of safety of the combination of drug dose with low energy localized light irradiation
Part I: Photosafety (sunburn) Testing | 1 month
  Determination of skin Minimal Erythema Dose (MED) following infusion of RM-1929
Part II: Maximum Tolerated Dose (MTD) or Maximum Feasible Dose (MFD) of a fixed drug dose with fixed light dose | 1 month
  Determination of MTD or MFD of fixed drug dose with fixed light dose
Part II: Safety with repeat dosing | 2 years or until death
  Safety parameters associated with repeat dosing

SECONDARY OUTCOMES:
Part I: Tumor response | 2 months
  Document tumor response using response assessment in solid tumors version 1.1 (RECIST 1.1), including additional assessment of target lesion volumetrics
Part 1: Tumor reduction/necrosis | 2 month
  Document tumor reduction/necrosis using Choi criteria
Part I: Pharmacokinetics of RM-1929 and for both RM-1929 and unconjugated IRDye 700DX (Cmax, T 1/2, AUC, CL and Vss) | 1 month
Part I: Immunogenic response to RM-1929 | 2 month
  To assess antibodies to RM-1929 or cetuximab
Part II: Tumor Response | 2 months
  Assessed using RECIST 1.1
Part II: Tumor Reduction | 2 months
  Evaluation by CT scans, clinical measurement, photographs, biopsies, symptom relief and ECOG performance
Part II: Immunogenic response to RM-1929 | 2 months
  To assess antibodies to RM-1929 or cetuximab

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Centura Health Research Center, Denver, Colorado
  - Rush University Cancer Center, Chicago, Illinois
  - Virginia Piper Cancer Institute, part of Allina Health System, Minneapolis, Minnesota
  - University of Oklahoma Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cognetti DM, Johnson JM, Curry JM, Kochuparambil ST, McDonald D, Mott F, Fidler MJ, Stenson K, Vasan NR, Razaq MA, Campana J, Ha P, Mann G, Ishida K, Garcia-Guzman M, Biel M, Gillenwater AM. Phase 1/2a, open-label, multicenter study of RM-1929 photoimmunotherapy in patients with locoregional, recurrent head and neck squamous cell carcinoma. Head Neck. 2021 Dec;43(12):3875-3887. doi: 10.1002/hed.26885. Epub 2021 Oct 9. PMID 34626024